CLINICAL TRIAL: NCT02467647
Title: Phase 1 Study of the Effects of Huang-Lian-Jie-Du-Tang（HLJDT) on the Survival of Patients With Multiple Myeloma in Maintain Therapy
Brief Title: The Effects of Huang-Lian-Jie-Du-Tang（HLJDT) on the Survival of Patients With Multiple Myeloma in Maintain Therapy
Acronym: HLJDT-2016
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan University (Other)
Collaborators: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Shangqin Liu, Professor, Wuhan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HLJDT-2016
Record Dates: First submitted 2013-06-15; First posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide; huang-lien-chieh-tu-tang

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Arm A: HLJDT 150ml three times per day for 6 months and Thalidomide 100mg once per day for 6 months
  Interventions: Drug: Thalidomide; Drug: HLJDT
- B (Active Comparator): Arm B: Thalidomide 100mg oral once per day for 6 months
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide
Drug: HLJDT
  Arms: A

SUMMARY:
To investigate the efficacy of the combination of Thalidomide and Huang-Lian-Jie-Du-Tang on the patients with multiple myeloma in maintain therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients can take HLJDT

Exclusion Criteria:

* patients can not take HLJDT

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival of patients with multiple myeloma treated with Huang-Lian-Jie-Du-Tang（HLJDT) in maintain therapy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shangqin Liu, PhD, Study Chair — Zhongnan Hospital
Locations (1):
- Wuhan University, Wuhan, Hubei, China

REFERENCES:
- [Background] Ma Z, Otsuyama K, Liu S, Abroun S, Ishikawa H, Tsuyama N, Obata M, Li FJ, Zheng X, Maki Y, Miyamoto K, Kawano MM. Baicalein, a component of Scutellaria radix from Huang-Lian-Jie-Du-Tang (HLJDT), leads to suppression of proliferation and induction of apoptosis in human myeloma cells. Blood. 2005 Apr 15;105(8):3312-8. doi: 10.1182/blood-2004-10-3915. Epub 2004 Dec 30. PMID 15626742
- [Background] Liu S, Ma Z, Cai H, Li Q, Rong W, Kawano M. Inhibitory effect of baicalein on IL-6-mediated signaling cascades in human myeloma cells. Eur J Haematol. 2010 Feb 1;84(2):137-44. doi: 10.1111/j.1600-0609.2009.01365.x. Epub 2009 Oct 28. PMID 19878271
- See also: Related Info — http://ubeliu.haodf.com